CLINICAL TRIAL: NCT01354808
Title: ACCELerated Inhibition of Platelet Aggregation, Inflammation and Ischemia-reperfusion Injury by Adjunctive Cilostazol Loading in Patients With Acute Coronary Syndrome
Brief Title: ACCEL-LOADING-ACS Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCEL-LOADING
Record Dates: First submitted 2011-05-15; First posted 2011-05-17 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Platelet Aggregation Inhibitors; Anti-inflammatory Agent; Myocardial Reperfusion Injury
Keywords: Cilostazol; Platelet; Inflammation; Myonecrosis
MeSH Terms: conditions — Myocardial Reperfusion Injury; Inflammation | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAPT (Active Comparator)
  Interventions: Drug: Dual Anti-Platelet Therapy (DAPT)
- TAPT (Experimental)
  Interventions: Drug: Triple Anti-Platelet Therapy (TAPT)

INTERVENTIONS:
Drug: Dual Anti-Platelet Therapy (DAPT) — * Loading: aspirin 300mg + clopidogrel 600mg
  * Maintenance: aspirin 200mg/d + clopidogrel 75mg/d for 1 month
  Arms: DAPT
Drug: Triple Anti-Platelet Therapy (TAPT) — * Loading: cilostazol 200mg + aspirin 300mg + clopidogrel 600mg
  * Maintenance: cilostazol 100mg bid+ aspirin 200mg/d+ clopidogrel 75mg/d for 1 month
  Arms: TAPT

SUMMARY:
The purpose of this study is to determine whether adjunctive cilostazol loading/maintenance to standard treatment (aspirin, clopidogrel, and statin) is effective in reduction of major adverse cardiovascular events, platelet activation, inflammation and myonecrosis in patients with non-ST-elevation acute coronary syndrome (ACS)undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
In ACS patients, platelet activation, inflammation, and ischemia-reperfusion injury can be closely associated with the risk of post-PCI myonecrosis and ischemic events occurrence. In the ACCEL-AMI (Adjunctive Cilostazol versus high maintenance-dose ClopidogrEL in patients with Acute Myocardial Infarction)study, adjunctive cilostazol increased platelet inhibition compared with double-dose clopidogrel. Meanwhile, statins can reduce the extent of myonecrosis via limiting inflammation and myocardial infarct size by activating phosphatidylinositol-3-kinase (PI3K), ecto-5'-nucleotidase, Akt/endothelial nitric oxide synthase (eNOS), and the downstream effectors inducible nitric oxide synthase (iNOS) and cyclooxygenase-2 (COX-2). Inhibition of PI3K, adenosine receptors, eNOS, iNOS, or COX-2 abrogates the protective effects of statins. In animal study, the combination of low-dose statin with cilostazol synergistically limits infarct size. Multiple studies have shown that cilostazol can influence inflammation and RISK pathway using the similar pathway with statin. This study will be performed to evaluate the role of adjunctive cilostazol in platelet inhibition, inflammation, and myonecrosis compared with standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* Non-ST-elevation ACS patients undergoing PCI within 48 hours after hospitalization

Exclusion Criteria:

* ST segment elevation acute myocardial infarction
* NSTE ACS with high-risk features warranting emergency coronary angiography
* Oral anticoagulation therapy with warfarin
* Use of pre-procedural glycoprotein IIb/IIIa inhibitor
* Contraindication to antiplatelet therapy
* AST or ALT ≥ 3 times upper normal
* Left ventricular ejection fraction < 30%
* WBC < 3,000/mm3, platelet < 100,000/mm3
* Creatinine ≥ 3 mg/dl
* stroke within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 1 month
  Composite of cardiac death, MI and ischemia-driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
P2Y12 reaction unit levels in the 2 arms | 1 month
MACE incidence according to P2Y12 reaction unit | 1 month
any post-procedural increase of markers of myocardial injury above ULN | 1 month
post-procedural variations from baseline of hs-CRP levels in the 2 arms | 1 month
ACUITY major/minor bleeding rate | 1 month
24hr post-procedural variations from baseline of inflammation markers (IL-6, TNF-alpha, cell adhesion molecules (VCAM, ICAM, E-selectin) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Kyounghoon Lee, MD, PhD, Principal Investigator — Gil hospital; Jae-Hyeong Park, MD, PhD, Principal Investigator — Chungnam National University Hospital; Keun-Ho Park, MD, Principal Investigator — Heart Center of Chonnam National University Hospital; Jon Suh, MD, PhD, Principal Investigator — Soon Chun Hyang University; Sang-Yong Yoo, MD, PhD, Principal Investigator — Gangneung Asan Medical Center
Locations (1):
- Gyeonsang National University Hospital, Jinju, Gyeonsangnam-do, South Korea

REFERENCES:
- [Result] Patti G, Pasceri V, Colonna G, Miglionico M, Fischetti D, Sardella G, Montinaro A, Di Sciascio G. Atorvastatin pretreatment improves outcomes in patients with acute coronary syndromes undergoing early percutaneous coronary intervention: results of the ARMYDA-ACS randomized trial. J Am Coll Cardiol. 2007 Mar 27;49(12):1272-8. doi: 10.1016/j.jacc.2007.02.025. PMID 17394957
- [Result] Jeong YH, Hwang JY, Kim IS, Park Y, Hwang SJ, Lee SW, Kwak CH, Park SW. Adding cilostazol to dual antiplatelet therapy achieves greater platelet inhibition than high maintenance dose clopidogrel in patients with acute myocardial infarction: Results of the adjunctive cilostazol versus high maintenance dose clopidogrel in patients with AMI (ACCEL-AMI) study. Circ Cardiovasc Interv. 2010 Feb 1;3(1):17-26. doi: 10.1161/CIRCINTERVENTIONS.109.880179. Epub 2010 Jan 26. PMID 20118150